CLINICAL TRIAL: NCT06464822
Title: Prospective Data-Collection for Assessment on Efficacy of Invasive Weight Management Program for Morbidly Obese Patients - IPSS and LUTS
Brief Title: Prospective Data on Bariatric Surgery Effect on IPSS and LUTS
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Alex Qinyang Liu, Medical Officer, Chinese University of Hong Kong
Other Study IDs: CREC 2008.497-T
Record Dates: First submitted 2024-06-07; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Bariatric Surgery Candidate; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: For patients decide not for bariatric surgery
- Intervention Group: For patient decided for Bariatric surgery
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — weight control procedures, including intragastric balloon (IGT) [5], laparoscopic adjustable gastric banding (LAGB) [6], laparoscopic gastric bypass (LGB) operation and laparoscopic sleeve gastrectomy (LSG)
  Groups: Intervention Group

SUMMARY:
To establish a central database on clinical parameters for patients who has morbid obesity, which aiming at

1. to compare the results of those with or without receiving invasive bariatric treatment in Prince of Wales Hospital ( Multidiciplinary Clinic of Metabolic & Bariatric Surgery) and CUHK Medical Centre (Weight Management & Metabolic Surgery Clinic).
2. To audit and compare outcome between PWH, CUHK Medical Centre, and with other bariatric surgery centers in Hong Kong (Hong Kong Bariatric & Metabolic Surgery Registry)
3. To compare outcome with the regional/international center databse for benchmarking performance of HK bariatric surgery

DETAILED DESCRIPTION:
Morbid obesity causes or exacerbates many diseases (DM, HT, sleep apnea, atherosclerosis etc) and is associated with major physical and psychosocial disability [1]. Moreover, ethnic background can also affect BMI-related disease risk as Southeast Asia populations have a higher risk of developing diabetes and cardiovascular disease than do Caucasian who have the same BMI values [2]. Non-surgical intervention, like diet and exercise plus augmented by drug therapy and behavioral modification, often provide an unsustainable and insufficient weight loss in morbidly obese patients (BMI > 40). The benefits of bariatric surgery is the effectiveness in achieving substantial (~50% excessive body weight loss) and sustainable weight control and improve co-morbidity and overall survival [3, 5, 4].

The Department of Surgery of CUHK is a pioneer in the development of bariatric surgery in Hong Kong. Since 2001, the investigators have introduced a variety of weight control procedures, including intragastric balloon (IGT) [5], laparoscopic adjustable gastric banding (LAGB) [6], laparoscopic gastric bypass (LGB) operation and laparoscopic sleeve gastrectomy (LSG) [7] in the region. Currently the investigators are holding the greatest volume of obesity cases and operative experience in this clinical subspecialty within Hong Kong. There is no comparable institution in HK as far as expertise in bariatric surgery's concerned. Since 2001, the investigators have received 510 referrals for bariatric surgery and have performed more than 220 operations thus far without mortality. The investigators foresee that the demand for such surgery is going to be huge in the future, especially in China. The number of cases treated reveals that the trend is on the increase. Furthermore, the Union Hospital has since inauguration been a working and training partner of the Faculty of Medicine, CUHK. In 2006, UH has established her weight management center and with the collaboration between her and CUHK, the investigators had established the Joint bariatric surgery research center in 2007. This collaboration provided us rooms for further development in the field of bariatric surgery.

Up till now, our initial results of previous prospective cohort received these procedures were promising without operative mortality. In a recent audit on our bariatric surgery service, the mean excessive weight loss for procedures LAGB, LSG and LGB were 34%, 51% and 61% at 2 years respectively [8]. In order to maintain the optimal outcome and seek for rooms of improvement, a proper data collection for both research and auditing (for PWH / CUHK MC / HK local audit & for bench marking with international standard) is necessary.

In order to extend our research and data collection for analysis, the investigators would like to set up a central database on patients who seeks for or received interventional bariatric procedures.

Objective To establish a central database on clinical parameters for patients who has morbid obesity, which aiming at

1. to compare the results of those with or without receiving invasive bariatric treatment in Prince of Wales Hospital ( Multidiciplinary Clinic of Metabolic & Bariatric Surgery) and CUHK Medical Centre (Weight Management & Metabolic Surgery Clinic).
2. To audit and compare outcome between PWH, CUHK Medical Centre, and with other bariatric surgery centers in Hong Kong (Hong Kong Bariatric & Metabolic Surgery Registry)
3. To compare outcome with the regional/international center databse for benchmarking performance of HK bariatric surgery

Study design Prospective cohort study

Sample size Since the current protocol is a prospective data collection of all bariatric surgical patients, the investigators estimate the yearly recruitment is approximately 200-250 patients. The investigators will not set limitation on the number of subjects recruited but will review this protocol every 5 years for necessary amendment and update.

ELIGIBILITY:
Inclusion Criteria

1. Patients with BMI >25
2. Patient who attended either the PWH Multidiciplinary Clinic of Metabolic & Bariatric Surgery to seek for treatment of severe obesity.
3. Consented patients (age >18).

Exclusion Criteria

1. Patient unable or unwilling to give written consent
2. Special population, e.g. prisoner, mentally disabled, investigators' student or employees.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who has morbid obesity and attended bariatric clinic of Prince of Wales Hospital
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
IPSS | Annually up to 10 years post-operatively
  International prostate symptom score
BMI | Annually up to 10 years post-operatively
  Body mass index
Percentage excess body weight loss | Annually up to 10 years post-operatively
  The amount of body mass lost due to bariatric surgery
Short Form Health Survey | Annually up to 10 years post-operatively
  SF 36
Eating Disorder Examination Questionnaire | Annually up to 10 years post-operatively
  EDE-Q
Adverse events | Up to 30 days post-operatively
  Side effect / new symptom after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data on individual participants and the study protocol will be available to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in an approved and methodologically sound proposal. Data requestors needing to sign a data access agreement.